CLINICAL TRIAL: NCT00894556
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Crossover Trial to Evaluate the Efficacy and Tolerability of Rizatriptan 10 mg for the Treatment of Acute Migraine in Sumatriptan Non-Responders
Brief Title: A Study to Evaluate the Efficacy and Tolerability of Rizatriptan for Treatment of Acute Migraine (0462-087)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0462-087; 2009_587
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Results first posted 2011-01-20 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2022-02

CONDITIONS: Acute Migraine
Keywords: Treatment of acute migraine with or without aura in adults
MeSH Terms: interventions — rizatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Sequence A (Experimental): Rizatriptan - Rizatriptan - Placebo
  Interventions: Drug: rizatriptan; Drug: Comparator: Placebo
- Treatment Sequence B (Experimental): Rizatriptan - Placebo - Rizatriptan
  Interventions: Drug: rizatriptan; Drug: Comparator: Placebo
- Treatment Sequence C (Experimental): Placebo - Rizatriptan - Rizatriptan
  Interventions: Drug: rizatriptan; Drug: Comparator: Placebo
- Baseline Phase (Other): Sumatriptan
  Interventions: Drug: Comparator: Sumatriptan

INTERVENTIONS:
Drug: rizatriptan — Single dose of 10 mg orally disintegrating tablet at onset of migraine attack
  Arms: Treatment Sequence A; Treatment Sequence B; Treatment Sequence C
Drug: Comparator: Placebo — Placebo to Rizatriptan
  Arms: Treatment Sequence A; Treatment Sequence B; Treatment Sequence C
Drug: Comparator: Sumatriptan — single dose of generic sumatriptan 100 mg at onset of migraine attack
  Arms: Baseline Phase

SUMMARY:
A study to provide evidence supporting the benefit of Rizatriptan in patients who have an inadequate response to sumatriptan.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a history of migraine with or without aura for 1 year or more with 2-8 moderate or severe migraine attacks per month
* Patient generally does not respond to treatment with sumatriptan
* Patient of reproductive potential agrees to remain abstinent or use one method of highly effective birth control (i.e. IUD, condoms, hormonal contraceptive, diaphragm, vasectomy) for the duration of the study
* Patient is able to complete paper diary

Exclusion Criteria:

* Patient is pregnant or breast feeding or excepts to become pregnant during the study
* Patient has history of mild migraine attacks or migraines that usually resolve spontaneously in less than 2 hours
* Patient has basilar or hemiplegic migraines
* Patient is unable to distinguish between migraine attacks from other types of headaches
* Patient has more than 15 headache-days per month
* Patient was greater than 50 years old at age of migraine onset
* Patient has failed to respond to 3 or more triptans
* Patient has a repeated history of failing to respond to or tolerate rizatriptan
* Patient uses opioids as primary migraine therapy
* Patient uses daily opioids
* Patient has a history of Cerebrovascular Accident (CVA) or other significant cardiovascular disease
* Patient has uncontrolled hypertension
* Patient has a history of neoplastic disease
* Patient is taking a serotonin reuptake inhibitor (SSRI or SNRI) where the dose has changed 3 months prior to screening
* Patient has a history of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-06-10 (Actual); Primary Completion 2010-01-12 (Actual); Study Completion 2010-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Seeburger JL, Taylor FR, Friedman D, Newman L, Ge Y, Zhang Y, Hustad CM, Lasorda J, Fan X, Hewitt D, Ho T, Connor KM. Efficacy and tolerability of rizatriptan for the treatment of acute migraine in sumatriptan non-responders. Cephalalgia. 2011 May;31(7):786-96. doi: 10.1177/0333102410390399. Epub 2010 Nov 15. PMID 21078681

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 21 study centers in the United States.
  First Patient In: 10-Jun-2009;
  First Patient Treated: 26-Jun-2009
  Last Patient Last Visit: 12-Jan-2010;
  Last Patient Treated: 25-Dec-2009
Pre-assignment Details: Participants who met entry criteria but had evidence of suicidality or were severely depressed (based on
  questionnaire scores) were excluded. Within 2 months of entry, participants were to treat a moderate/
  severe migraine attack with sumatriptan 100 mg and were randomized if they still had moderate or severe
  pain at 2 hours post-dose.
Groups:
- Rizatriptan / Rizatriptan / Placebo: Each patient was randomized to receive one of 3 treatment sequences. Three qualifying migraines were
  then treated based on the prescribed sequence. Two migraine attacks were treated with rizatriptan and one
  with placebo.
  The first migraine was treated with Rizatriptan 10 mg Orally Disintegrating Tablet (ODT); the second migraine with Rizatriptan 10 mg ODT; the third migraine with placebo.
- Rizatriptan / Placebo / Rizatriptan: Each patient was randomized to receive one of 3 treatment sequences. Three qualifying migraines were
  then treated based on the prescribed sequence. Two migraine attacks were treated with rizatriptan and one
  with placebo.
  The first migraine was treated with Rizatriptan 10 mg ODT; the second migraine with placebo; and the third migraine with Rizatriptan 10 mg ODT.
- Placebo / Rizatriptan / Rizatriptan: Each patient was randomized to receive one of 3 treatment sequences. Three qualifying migraines were
  then treated based on the prescribed sequence. Two migraine attacks were treated with rizatriptan and one
  with placebo.
  The first migraine was treated with Placebo; the second migraine with Rizatriptan 10mg ODT; and the third migraine with Rizatriptan 10 mg ODT
- Sumatriptan 100 mg: Pre-Randomization Phase conducted 2 months prior to Study Randomization. Eligible participants were to treat a moderate/severe migraine attack with sumatriptan 100 mg. Those who failed to respond to sumatriptan (i.e. continued to experience moderate or severe pain at 2 hours post dose) were classified as non-responders and were entered into the double-blind treatment phase of the study.
Period: Baseline Phase
Arm/Group | Rizatriptan / Rizatriptan / Placebo | Rizatriptan / Placebo / Rizatriptan | Placebo / Rizatriptan / Rizatriptan | Sumatriptan 100 mg
Started | 0 | 0 | 0 | 194
Completed | 0 | 0 | 0 | 109
Not Completed | 0 | 0 | 0 | 85
Not completed — Did not meet Randomization Criteria | 0 | 0 | 0 | 85
Period: Treatment Phase
Arm/Group | Rizatriptan / Rizatriptan / Placebo | Rizatriptan / Placebo / Rizatriptan | Placebo / Rizatriptan / Rizatriptan | Sumatriptan 100 mg
Started | 37 (Participants who were randomized into the treatment phase) | 36 (Participants who were randomized into the treatment phase) | 36 (Participants who were randomized into the treatment phase) | 0
Completed | 33 (Participants who treated 3 acute migraine attacks with study medication during the treatment phase) | 32 (Participants who treated 3 acute migraine attacks with study medication during the treatment phase) | 35 (Participants who treated 3 acute migraine attacks with study medication during the treatment phase) | 0
Not Completed | 4 | 4 | 1 | 0
Not completed — Lost to Follow-up | 2 | 3 | 1 | 0
Not completed — Lack of Qualifying Event | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rizatriptan / Rizatriptan / Placebo: The first migraine was treated with Rizatriptan 10 mg Orally Disintegrating Tablet (ODT); the second migraine with Rizatriptan 10 mg ODT; the third migraine with placebo.
- Rizatriptan / Placebo / Rizatriptan: The first migraine was treated with Rizatriptan 10 mg ODT; the second migraine with placebo; and the third migraine with Rizatriptan 10 mg ODT.
- Placebo / Rizatriptan / Rizatriptan: The first migraine was treated with Placebo; the second migraine with Rizatriptan 10mg ODT; and the third migraine with Rizatriptan 10 mg ODT
- Total: Total of all reporting groups
Arm/Group | Rizatriptan / Rizatriptan / Placebo | Rizatriptan / Placebo / Rizatriptan | Placebo / Rizatriptan / Rizatriptan | Total
Number analyzed (Participants) | 37 | 36 | 36 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (13.4) | 43.6 (8.9) | 43.5 (10.2) | 43.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 30 | 95
  Male | 5 | 3 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 6
  Not Hispanic or Latino | 34 | 35 | 34 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 3 | 11
  White | 31 | 31 | 30 | 92
  More than one race | 2 | 1 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief (PR)
Description: Pain severity was rated by the participants in a paper diary. Pain severity rating scale: 0 (no pain), 1 (mild pain), 2 (moderate pain), or 3 (severe pain). Pain relief (PR) is defined as a reduction in headache severity from Grade 3/2 at baseline to Grade 1/0 post dose.
Time Frame: 2 hours post dose
Population: The FAS population included all randomized participants who had at least one evaluable attack. To be considered an evaluable attack the participant must have administered study treatment for this attack and must have had both a baseline severity measurement and at least one post-dose efficacy measurement prior to or including the 2-hour time point.
Measure: Number; unit: attacks
Units Other Than Participants: Evaluable Attacks
Groups:
- Rizatriptan: Migraines were treated with Rizatriptan 10 mg ODT.
  Although a patient may have appeared twice in the rizatriptan group, the patient was counted only once for the rizatriptan group. It is possible for one patient to be counted in both the rizatriptan and placebo groups.
- Placebo: Migraines were treated with placebo
Arm/Group | Rizatriptan | Placebo
Number analyzed (Participants) | 102 | 99
Number analyzed (Evaluable Attacks) | 202 | 99
attacks
  Resulting in PR at 2 hours post dose | 102 | 21
  Not resulting in PR at 2 hours post dose | 100 | 78
Statistical Analysis 1: Comparison: Rizatriptan vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized Linear Mixed Model (GLIMMIX); An unstructured covariance matrix was used to model the correlation among repeated measurements within patient

2. Secondary Outcome: Pain Freedom (PF)
Description: Headache pain severity, relative to the administration of study medication, was rated by the participants in a paper diary. Pain severity rating scale: 0 (no pain), 1 (mild pain), 2 (moderate pain), or 3 (severe pain). Pain freedom (PF) is defined as a reduction in headache severity from Grade 3/2 at baseline to Grade 0 (no pain) post dose.
Time Frame: 2 hours post dose
Population: as for outcome 1
Measure: Number; unit: attacks
Units Other Than Participants: Evaluable Attacks
Arm/Group | Rizatriptan | Placebo
Number analyzed (Participants) | 102 | 99
Number analyzed (Evaluable Attacks) | 202 | 99
attacks
  Resulting in PF at 2 hours post dose | 46 | 12
  Not resulting in PF at 2 hours post dose | 156 | 87
Statistical Analysis 1: Comparison: Rizatriptan vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized Linear Mixed Model (GLIMMIX); An unstructured covariance matrix was used to model the correlation among repeated measurements within patient

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time that participants were enrolled (signed informed consent) through 14 days after the last dose of study medication.
Description: Participants reported adverse events in a paper diary and were collected by the site at Visits 2 and 3, and 14 days after the last dose of study medication. AEs that occurred in the Baseline Phase (prior to randomization) are reported as a separate arm. Events not applicable to a particular Study Phase are reported as (0/0).
Groups:
- Rizatriptan 10 mg: Patients took at least one dose of study medication. It is possible for one patient to be counted twice (once in each treatment group).
  Although a patient may have had two or more adverse events of the same type, the patient is counted only once for that type of adverse event.
  Adverse events occurring within 14 days of administration of Rizatriptan 10 mg are attributed to Rizatriptan 10 mg group even if placebo was administered more recently.
- Sumatriptan 100 mg: Adverse Events that occurred in the Baseline Phase (prior to taking study medication) are identified in the tables as "Baseline Phase"
Arm/Group | Rizatriptan 10 mg | Placebo | Sumatriptan 100 mg
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/100 | 0/194
Other Adverse Events (participants affected / at risk) | 18/102 | 3/100 | 29/194
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Rizatriptan 10 mg (N=102) | Placebo (N=100) | Sumatriptan 100 mg (N=194)
Tachycardia - Baseline Phase (Cardiac disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Motion Sickness - Baseline Phase (Ear and labyrinth disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Eyelid Pain - Baseline Phase (Eye disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Abdominal pain - Baseline Phase (Gastrointestinal disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Abdominal pain upper - Baseline Phase (Gastrointestinal disorders) | 0/0 | 0/0 | 2 — Pre-Randomization reported Adverse Event
Dry mouth - Baseline Phase (Gastrointestinal disorders) | 0/0 | 0/0 | 2 — Pre-Randomization reported Adverse Event
Nausea - Baseline Phase (Gastrointestinal disorders) | 0/0 | 0/0 | 4 — Pre-Randomization reported Adverse Event
Paraesthesia oral - Baseline Phase (Gastrointestinal disorders) | 0/0 | 0/0 | 2 — Pre-Randomization reported Adverse Event
Asthenia - Baseline Phase (General disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Chest discomfort - Baseline Phase (General disorders) | 0/0 | 0/0 | 3 — Pre-Randomization reported Adverse Event
Fatigue - Baseline Phase (General disorders) | 0/0 | 0/0 | 2 — Pre-Randomization reported Adverse Event
Oedema peripheral - Baseline Phase (General disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Pain - Baseline Phase (General disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Hordeolum - Baseline Phase (Infections and infestations) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Nasopharyngitis - Baseline Phase (Infections and infestations) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Rhinitis - Baseline Phase (Infections and infestations) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Foot fracture - Baseline Phase (Injury, poisoning and procedural complications) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Heart rate increased - Baseline Phase (Investigations) | 0/0 | 0/0 | 2 — Pre-Randomization reported Adverse Event
Back pain - Baseline Phase (Musculoskeletal and connective tissue disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Muscle spasms - Baseline Phase (Musculoskeletal and connective tissue disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Muscle tightness - Baseline Phase (Musculoskeletal and connective tissue disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Neck pain - Baseline Phase (Musculoskeletal and connective tissue disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Cognitive disorder - Baseline Phase (Nervous system disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Dizziness - Baseline Phase (Nervous system disorders) | 0/0 | 0/0 | 9 — Pre-Randomization reported Adverse Event
Headache - Baseline Phase (Nervous system disorders) | 0/0 | 0/0 | 3 — Pre-Randomization reported Adverse Event
Migraine - Baseline Phase (Nervous system disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Paraesthesia - Baseline Phase (Nervous system disorders) | 0/0 | 0/0 | 3 — Pre-Randomization reported Adverse Event
Sinus headache - Baseline Phase (Nervous system disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Anxiety - Baseline Phase (Psychiatric disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Insomnia - Baseline Phase (Psychiatric disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Metrorrhagia - Baseline Phase (Reproductive system and breast disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Dyspnoea - Baseline Phase (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Throat tightness - Baseline Phase (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/0 | 2 — Pre-Randomization reported Adverse Event
Hot flush - Baseline Phase (Vascular disorders) | 0/0 | 0/0 | 1 — Pre-Randomization reported Adverse Event
Eyelid ptosis - Treatment Phase (Eye disorders) | 0 | 1 | 0/0 — Post-Randomization reported Adverse Event
Vision blurred - Treatment Phase (Eye disorders) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Abdominal pain upper - Treatment Phase (Gastrointestinal disorders) | 2 | 1 | 0/0 — Post-Randomization reported Adverse Event
Diarrhoea - Treatment Phase (Gastrointestinal disorders) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Nausea - Treatment Phase (Gastrointestinal disorders) | 4 | 0 | 0/0 — Post-Randomization reported Adverse Event
Fatigue - Treatment Phase (General disorders) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Feeling of relaxation - Treatment Phase (General disorders) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Gait disturbance - Treatment Phase (General disorders) | 0 | 1 | 0/0 — Post-Randomization reported Adverse Event
Influenza like illness - Treatment Phase (General disorders) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Sensation of pressure - Treatment Phase (General disorders) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Facial bones fracture - Treatment Phase (Injury, poisoning and procedural complications) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Wrist fracture - Treatment Phase (Injury, poisoning and procedural complications) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Myokymia - Treatment Phase (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Melanocytic naevus - Treatment Phase (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Cognitive disorder - Treatment Phase (Nervous system disorders) | 0 | 1 | 0/0 — Post-Randomization reported Adverse Event
Dizziness - Treatment Phase (Nervous system disorders) | 4 | 1 | 0/0 — Post-Randomization reported Adverse Event
Dysgeusia - Treatment Phase (Nervous system disorders) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Paraesthesia - Treatment Phase (Nervous system disorders) | 2 | 1 | 0/0 — Post-Randomization reported Adverse Event
Sinus headache - Treatment Phase (Nervous system disorders) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Somnolence - Treatment Phase (Nervous system disorders) | 2 | 0 | 0/0 — Post-Randomization reported Adverse Event
Syncope - Treatment Phase (Nervous system disorders) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Insomnia - Treatment Phase (Nervous system disorders) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event
Hot flush - Treatment Phase (Vascular disorders) | 1 | 0 | 0/0 — Post-Randomization reported Adverse Event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.